CLINICAL TRIAL: NCT07324343
Title: Which Patient Group Shows Greater Improvement With Patient Education Alone in Rotator Cuff-Related Shoulder Pain? - A Cohort Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve Koyuncu Cenikli, Research Asistant, PT, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2150061
Record Dates: First submitted 2025-11-27; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain Syndrome; Subacromial Pain Syndrome; Rotator Cuff Related Shoulder Pain; Patient Education
Keywords: patient education; Rotator Cuff Related Shoulder Pain
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Education (Experimental): Participants in this study will receive structured patient education sessions for rotator cuff-related shoulder pain.
  Interventions: Behavioral: Questionnaire Validation; Behavioral: Patient Education

INTERVENTIONS:
Behavioral: Questionnaire Validation — During the Turkish adaptation of the PKQ-RCRSP questionnaire, written permission was obtained from the original developer. At least two experts independently translated the questionnaire into Turkish, and a single reconciled version was created. This version was back-translated by an independent translator to ensure semantic and conceptual equivalence. Revisions were made following expert panel review and pilot testing.
  For validation, the PKQ-RCRSP will be administered to participants at baseline (V0). One week later (V1), the questionnaire will be repeated, and participants will be asked if their shoulder problem or knowledge has significantly changed in the past week. Those answering "Yes," who do not return, or who receive any intervention will be excluded from the test-retest analysis. Results from participants answering "No" will complete the test-retest analysis, and all participants' data will be included in other validity analyses. This concludes the validation phase.
Behavioral: Patient Education — Participants in this arm will receive structured patient education sessions for rotator cuff-related shoulder pain. The program consists of two 30-minute face-to-face sessions delivered by a physiotherapist with at least 5 years of experience in orthopedic rehabilitation. Educational topics include disease information, symptom management, treatment options, reducing fear of movement, exercise promotion, pain and stress management, physical activity recommendations, nutrition advice, and lifestyle-specific guidance. Informational brochures will be provided after the first session. The second session, delivered two weeks later, focuses on reviewing progress and enhancing motivation; no new information will be provided.

SUMMARY:
The primary aim of this study is to determine the clinical effectiveness of patient education alone in individuals with rotator cuff-related shoulder pain and to identify which patient subgroups benefit more from this approach. In addition, the translation and cultural adaptation of the "Patient Knowledge Questionnaire (PKQ-RCRSP)" into Turkish will be carried out to measure the level of patient knowledge regarding patient education.

DETAILED DESCRIPTION:
Individuals who present with shoulder pain to the Orthopedics and Traumatology Department, Shoulder-Elbow Surgery Outpatient Clinic of Göztepe Prof. Dr. Süleyman Yalçın City Hospital and who volunteer to participate will be included in our study. Before beginning the study, the purpose of the study will be explained to the participants, and all information regarding the study will be provided both verbally and in writing. Informed consent will be obtained from participants, confirming that they voluntarily agree to take part in the study. A total of 116 participants will be included in the study, and the PKQ-RCRSP questionnaire will be administered at baseline and after one week. Following the validation process, participants will receive two face-to-face patient education sessions. After the first patient education session, pain will be assessed at the 4th, 12th, and 24th week follow-ups using the Numerical Pain Rating Scale (NPRS); functional limitation will be assessed using the Shoulder Pain and Disability Index (SPADI); clinical improvement using the Global Rating of Change Scale (GRC); illness perception using the Brief Illness Perception Questionnaire (B-IPQ); patient knowledge level using the PKQ-RCRSP; health literacy using the European Health Literacy Survey-Short Form (HLS-EU-Q6); and physical activity level using the International Physical Activity Questionnaire (IPAQ).

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 years
* Shoulder pain persisting for at least 4 weeks
* Diagnosed by an orthopedic physician with impingement, subacromial bursitis, rotator cuff (RC) tendinopathy, or partial tear
* Activity-related pain ≥3 on the NPRS
* Cognitively able to understand the education and provide written informed consent

Exclusion Criteria:

* History of shoulder surgery
* Diagnosis of frozen shoulder, full-thickness or massive rotator cuff (RC) tear, or instability
* Presence of neurological or psychiatric conditions that prevent exercise
* History of physical therapy-rehabilitation or injection treatment within the past 6 months
* Pain persisting for more than 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | İmmediately before the first education session, and at 4 weeks, 12 weeks, and 24 weeks after the start of the education program.
  Pain intensity assessed using the Numerical Pain Rating Scale (NPRS).

SECONDARY OUTCOMES:
Patient Knowledge Questionnaire (PKQ-RCRSP) | Baseline, immediately before the first education session, and at 4 weeks, 12 weeks, and 24 weeks after the start of the education program.
  Patient knowledge regarding rotator cuff-related shoulder pain assessed

OTHER OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline, and at 4 weeks, 12 weeks, and 24 weeks after the start of the education program.
  Shoulder pain and functional disability assessed using the Shoulder Pain and Disability Index (SPADI).
Sociodemographic Characteristics | Baseline.
  Sociodemographic characteristics including age, sex, education level, occupation, and other relevant demographic variables collected using a Sociodemographic Assessment Form.
Patient-Reported Global Change Assessed by the Global Rating of Change Scale (GRC) | 4 weeks, 12 weeks, and 24 weeks after the start of the education program
  Patient-perceived overall change in condition assessed using the Global Rating of Change Scale (GRC).
Illness Perceptions Assessed by the Brief Illness Perception Questionnaire (B-IPQ) | Baseline and at 4 weeks, 12 weeks, and 24 weeks after the start of the education program.
  Patient perceptions of illness assessed using the Brief Illness Perception Questionnaire (B-IPQ).
European Health Literacy Survey - Short Form (HLS-EU-Q6) | Baseline, and at 4 weeks, 12 weeks, and 24 weeks after the start of the education program.
  Health literacy level assessed using the European Health Literacy Survey - Short Form (HLS-EU-Q6).
European Health Literacy Survey - Short Form (HLS-EU-Q6). | Baseline and at 12 weeks and 24 weeks after the start of the education program.
  Health literacy level assessed using the European Health Literacy Survey - Short Form (HLS-EU-
International Physical Activity Questionnaire - Short Form (IPAQ-SF / UFAA-KF) | Baseline and at 12 weeks and 24 weeks after the start of the education program.
  Physical activity level assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF).

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University Cerrahpasa Faculty of Health Sciences, İstanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No